CLINICAL TRIAL: NCT00541203
Title: Cardiac Computed Tomography In the Management of Patients With indeterminAte or inConclusive Stress Tests
Acronym: CT-MPACT
Status: Completed | Type: Observational
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Kavitha Chinnaiyan, Director, Cardiovascular Imaging Education, Corewell Health East
Other Study IDs: 2007-120
Record Dates: First submitted 2007-10-09; First posted 2007-10-10 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Coronary Disease
Keywords: tomography; coronary artery disease; Stress Test; Coronary Angiography
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Coronary CT angiography (CCTA) offers great promise as a risk stratification tool in patients with suspected CAD. It has been demonstrated in a multitude of accuracy studies to have a negative predictive value averaging over 95%. This leads to the hypothesis that a negative CCTA may preclude the need for invasive testing. The purpose of this randomized controlled study is to prospectively evaluate the role of CCTA on the management of patients with inconclusive or indeterminate stress test results.CCTA is able to provide not only information on presence and extent of coronary artery calcification, but detailed coronary anatomy as well.

SPECIFIC AIM # 1: To evaluate the diagnostic and prognostic performance of CCTA in patients with equivocal / intermediate stress test results as compared to conventional invasive coronary angiography.

SPECIFIC AIM # 2: To evaluate the utility of CCTA in prediction of major adverse cardiac events (MACE) compared to invasive coronary angiography at 30 days, 1 year, 3 years and 5 years.

DETAILED DESCRIPTION:
Outpatients scheduled to undergo cardiac catheterization and coronary angiography for the specific indication of inconclusive or indeterminate stress tests will be considered for this study. Patients will be initially screened by their cardiologist for the presence of inclusion/exclusion criteria, as well as pre-test and post-test likelihood of CAD.16, 17 All patients must have undergone a stress (exercise or pharmacologic) test within the past 3 months.

After consent, patients will be randomized 1:1 to undergo CCTA or cardiac catheterization. The decision whether or not to proceed with subsequent invasive cardiac catheterization (CCTA arm) or revascularization (catheterization arm) will be made by the patient's primary and interventional cardiologists respectively.

Inclusion:

1. Chest pain or other symptoms suggestive of coronary artery disease.
2. Pharmacologic/exercise stress test with SPECT (nuclear myocardial-heart perfusion imaging) within the past 3 months.
3. "Discordant or conflicting findings" clinical and stress results as outlined above.
4. Scheduled to undergo cardiac catheterization.
5. Able to provide informed consent.
6. Age equal to or greater than 18 years.

Exclusion:

1. Presence of pre-existing heart disease (prior heart attack, prior angiographic evidence of significant heart disease, prior heart surgery) or cardiomyopathy (ejection fraction less than or equal to 45%)
2. History of high blood pressure with severe left ventricular hypertrophy (thicken heart muscle), history of cor pulmonale (right heart chamber failure due to elevated blood pressures in the arteries delivering blood to the lungs).
3. Kidney insufficiency (creatinine greater than or equal to 1.6) or kidney failure requiring dialysis.
4. Inability or refusal to provide informed consent.
5. Psychological unsuitability or extreme claustrophobia (fear of closed in spaces).
6. Pregnancy or unknown pregnancy status.
7. Age less than 18 years.
8. Patients with known allergy to iodinated contrast, unable to tolerate pre-medication.
9. Inability to tolerate beta-blockers (medication to slow the heart rate), including those with COPD or asthma requiring maintenance inhaled bronchodilators or steroids, complete heart block, second-degree atrioventricular block.
10. Computed tomography imaging, or contrast administration, within the past 48 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Chest pain or other symptoms suggestive of coronary artery disease.
2. Pharmacologic/exercise stress test with SPECT within the past 3 months.
3. "Discordant" clinical and stress results as outlined above.
4. Scheduled to undergo cardiac catheterization.
5. Able to provide informed consent.
6. Age equal to or greater than 18 years.

Exclusion Criteria:

1. Presence of pre-existing CAD (prior myocardial infarction, prior angiographic evidence of significant coronary artery disease, prior coronary bypass surgery) or cardiomyopathy (ejection fraction < 45%)
2. History of hypertension with severe left ventricular hypertrophy, history of cor pulmonale.
3. Renal insufficiency (creatinine ≥1.6) or renal failure requiring dialysis.
4. Inability or refusal to provide informed consent.
5. Psychological unsuitability or extreme claustrophobia.
6. Pregnancy or unknown pregnancy status.
7. Age less than 18 years.
8. Patients with known allergy to iodinated contrast, unable to tolerate pre-medication.
9. Inability to tolerate beta-blockers, including those with COPD or asthma requiring maintenance inhaled bronchodilators or steroids, complete heart block, second-degree atrioventricular block.
10. Computed tomography imaging, or contrast administration, within the past 48 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers over 18 years of age; both genders; referred from participating cardiologist's offices
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kavitha Chinnaiyan, MD, Principal Investigator — Corewell Health East; Gilbert Raff, MD, Study Director — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States